CLINICAL TRIAL: NCT00714597
Title: A Multinational, Multicenter, Randomized, Double-Blind Study Comparing the Efficacy and Safety of AVE5026 With Enoxaparin for the Primary Prevention of Venous Thromboembolism in Acutely Ill Medical Patients With Restricted Mobility
Brief Title: Evaluation of AVE5026 in the Prevention of Venous Thromboembolism in Acutely Ill Medical Patients With Restricted Mobility
Acronym: SAVE-VEMED
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC10572; 2008-000228-13 (EudraCT Number)
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Venous Thromboembolism
Keywords: Venous thrombosis; Primary prevention
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — AVE 5026; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semuloparin (Experimental): Semuloparin sodium 20 mg (10 mg if Severe Renal Impairment [SRI]) once daily for 10-14 days
  Interventions: Drug: Semuloparin sodium
- Enoxaparin (Active Comparator): Enoxaparin sodium 40 mg (20 mg if Severe Renal Impairment [SRI]) once daily for 10-14 days
  Interventions: Drug: Enoxaparin sodium

INTERVENTIONS:
Drug: Semuloparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: AVE5026
  Arms: Semuloparin
Drug: Enoxaparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: Lovenox®
  Arms: Enoxaparin

SUMMARY:
The primary objective was to compare the efficacy of once daily [q.d] subcutaneous [s.c.] injections of Semuloparin sodium (AVE5026) with q.d. s.c. injections of Enoxaparin for the primary prevention of Venous Thromboembolic Events [VTE] in patients hospitalized for acute medical illness.

The secondary objectives were to evaluate the safety of AVE5026 and to document AVE5026 exposure in this population.

DETAILED DESCRIPTION:
Randomization had to take place just prior to the first study drug injection.

The total duration of observation per participant was 35-42 days from randomization broken down as follows:

* 10 to 14-day double-blind treatment period;
* 25 to 32-day follow-up period.

Mandatory bilateral compression ultrasound [CUS] had to be performed between 10 to 15 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

Patient with an acute medical condition requiring bed rest for at least 3 days, and hospitalized for at least one of the following medical conditions:

* Congestive heart failure (New York Heart Association [NYHA] class III/IV);
* Acute respiratory failure (not requiring mechanical ventilation);
* Acute infection (without septic shock)*;
* Acute rheumatic disorder*;
* Acute episode of inflammatory bowel disease*.

  * Patient with one of these conditions should have at least one additional risk factor for venous thromboembolism (VTE) among the following:

    * Age ≥ 75 years;
    * Active cancer or myeloproliferative disorders (having received treatment for cancer within the last 6 months);
    * Previous VTE;
    * Obesity;
    * Oral hormone therapy (antiandrogen or estrogen);
    * Chronic heart failure;
    * Chronic respiratory failure.

Exclusion Criteria:

* Previous surgery with general anesthesia within 30 days before inclusion in the study;
* Patient requiring a curative anticoagulant or thrombolytic treatment;
* Patient at risk of bleeding;
* Stroke;
* Known hypersensitivity to heparin or enoxaparin sodium;
* End stage renal disease or patient on dialysis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced Venous Thromboembolism Event (VTE) or VTE-related Death | From randomization up to 15 days after randomization or the day of the mandatory Compression Ultrasound (CUS), whichever came first
  VTE included:
  * asymptomatic proximal Deep Vein Thrombosis (DVT) detected by the mandatory CUS and confirmed by a Compression Ultrasound Adjudication Committee (CUSAC) after central and blind review of the mandatory CUS;
  * symptomatic DVT and non-fatal Pulmonary Embolism (PE) reported by the investigator and confirmed by a Central Independent Adjudication Committee (CIAC) after central and blind review of diagnosis tests.
  VTE-related Death included fatal PE and unexplained deaths.

SECONDARY OUTCOMES:
Percentage of Participants Who Experienced asymptomatic proximal DVT | From randomization up to 15 days after randomization or the day of the mandatory CUS, whichever came first.
Percentage of Participants Who Experienced Clinically Relevant Bleedings | From 1st study drug injection up to 3 days after last study drug injection
  Bleedings were centrally and blindly reviewed by the CIAC and classified as:
  * "major" (fatal, symptomatic in a critical area/organ, causing a post-operative drop in hemoglobin ≥2 g/dL or requiring post-operative transfusion ≥2 units of blood);
  * "clinically relevant non-major" (overt bleeding requiring medical intervention and not meeting criteria for major bleeding);
  * "Non-clinically relevant bleeding".
Percentage of Participants Who Required the Initiation of Curative Anticoagulant or Thrombolytic Treatment After VTE Assessment | From randomization up to 15 days after randomization or the day of mandatory CUS, whichever came first
  Initiation of curative anticoagulant or thrombolytic treatment after VTE assessment was defined from investigator's answer to the question "was the subject treated for VTE?" asked after the diagnostic tests for suspected VTE and after the mandatory CUS.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mismetti, MD, Principal Investigator — University Hospital of Saint-Etienne, France; Alexander Turpie, MD, Study Chair — HHS-General Hospital, Hamilton, Canada
Locations (22):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Riga, Latvia
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Auckland, New Zealand
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom